CLINICAL TRIAL: NCT06996795
Title: Investigating the Effects of Music Therapy on Sensory Processing, Adaptive Behavior and Social Interaction in Children With Autism
Brief Title: Effects of Music Therapy on Sensory Processing, Adaptive Behavior and Social Interaction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Kaya Ozturk, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HÜ-OT-LKO-05
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Music Therapy
Keywords: autism; sensory integration; music therapy; sensory processing; social interaction
MeSH Terms: conditions — Autistic Disorder | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Two groups with an intervention group and a control group
Who Masked: Outcomes Assessor
Masking Description: The therapist who conducted the assessment tests was unaware of the participants' group assignments (interventon or control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensory integration training and music therapy (Active Comparator): The intervention group will receive both sensory integration training and music therapy. Sensory integration will include sensory modulation activities, vestibular, proprioceptive, tactile, visual and auditory sensory studies. Music therapy will be applied with drums, maracas, cymbals and orf instruments. It will consist of body rhythms, breathing exercises and rhythm studies.
  Interventions: Behavioral: music therapy; Behavioral: sensory integration
- sensory integration training (Active Comparator): The control group will receive sensory integration training. Sensory integration will include sensory modulation activities, vestibular, proprioceptive, tactile, visual and auditory sensory studies.
  Interventions: Behavioral: sensory integration

INTERVENTIONS:
Behavioral: music therapy — Music therapy will be applied with drums, maracas, cymbals and orf instruments. It will consist of body rhythms, breathing exercises and rhythm studies.
  Arms: sensory integration training and music therapy
Behavioral: sensory integration — Sensory integration will include sensory modulation activities, vestibular, proprioceptive, tactile, visual and auditory sensory studies.

SUMMARY:
The purpose of our study is to examine the effects of music therapy on sensory processing, adaptive behavior, and social interaction in individuals with autism.

DETAILED DESCRIPTION:
The study was designed as a randomized controlled trial. A simple randomization method will be used to randomly assign individuals to two groups (intervention and control groups). A simple randomization method will be used where the intervention and control group papers are selected from a sealed envelope. Following the initial assessment of each participant, one of the papers labeled "intervention" or "control" will be randomly selected. This decision will determine whether the individual will be assigned to the intervention or control group. The study will be conducted at Hacettepe University. The study group and the control group will receive sensory integration training for 45 minutes per day, 2 days per week, for 6 weeks. The children in the control group will receive only sensory integration training, while the study group will receive music therapy training for 30 minutes per day, 2 days per week, for 6 weeks in addition to sensory integration training. Sociodemographic information of the children will be collected before the research and sensory processing problems of the children will be assessed with the Sensory Profile and adaptive behavioral skills will be assessed with the Adaptive Behavior Scale (ADS).

ELIGIBILITY:
Inclusion Criteria:

Having been diagnosed with autism spectrum disorder (ASD) by a child psychiatrist Being between the ages of 6-10 being able to cooperate

Exclusion Criteria:

Having any neurological, orthopedic or psychiatric diagnosis in addition to autism diagnosis Having undergone any surgical intervention in the last 3 months Being inadequate in understanding visual and auditory commands Having a visual and hearing impairment recorded in the health report

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
sensory profile | 1 month
  Sensory Profile: This assessment tool is used to determine the sensory profiles of children between the ages of 3-10. The test consists of 125 questions and a parent/caregiver with whom the child has one-on-one communication in his/her daily life answers the test questions. The test consists of three main sections: sensory processing, modulation and behavioral and emotional responses. The subsections of each main section consist of a total of 14 sections and 125 questions. The test takes approximately 30 minutes to administer. You are asked to mark one of the options: always, often, sometimes, occasionally and never. The assessment results are found by scoring from 1 to 5, giving 5 points to "never" and 1 point to "always". In this assessment, 1 point reflects a situation where there is a disordered behavior related to the sensory profile and 5 points reflects a situation where there is normal behavior. The Turkish adaptation of this test was made.

SECONDARY OUTCOMES:
Adaptive Behavior Scale | 1 month
  Adaptive Behavior Scale (ABS): The scale evaluates the child's adaptive behavior according to two basic criteria: the person's possession of basic skills such as self-care and personal hygiene, and avoiding behaviors that are not accepted by the environment, such as harming others and using physical violence. The Turkish validity study of the Adaptive Behavior Scale was conducted. The Adaptive Behavior Scale consists of two sections. The first section evaluates the skills and habits in nine behavioral areas that are important for the individual's development of independence in daily life. The second section is designed to measure non-adaptive behavior related to personality and behavioral disorders. If the behavior occurs "occasionally", "1" is marked, and if it occurs "frequently", "2" is marked. 25-30 minutes is considered sufficient for the application of the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No